CLINICAL TRIAL: NCT01877174
Title: MICHI™ Neuroprotection System (NPS+f) Filter Debris Analysis Study (The F-1 Study)
Status: Completed | Type: Observational
Sponsor: Silk Road Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: SRM-2013-01
Record Dates: First submitted 2013-05-27; First posted 2013-06-13 (Estimated); Last update posted 2014-09-03 (Estimated); Status verified 2014-09

CONDITIONS: Internal Carotid Artery Stenosis
Keywords: Internal Carotid Stenosis; Reverse Flow; Carotid stenting; MICHI(TM) NPS+f
MeSH Terms: conditions — Carotid Stenosis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The inline filter of the MICHI(TM) NPS+f System may contain debris that is released from the lesion during carotid stenting. It is the objective of the study to determine the volume and characteristics of the debris.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- MICHI(TM) NPS+f: Patients routinely treated with the CE marked MICHI(TM) NPS+f System
  Interventions: Device: MICHI(TM) NPS+f; Procedure: transcarotid stenting

INTERVENTIONS:
Device: MICHI(TM) NPS+f — Transcarotid delivery system for carotid stents with flow reversal
Procedure: transcarotid stenting

SUMMARY:
This study will be conducted in up to 10 hospitals in Europe, up to 75 patients will be enrolled. The purpose of the study is to evaluate any debris that may be captured in the inline filter of the MICHI(TM) Neuroprotection System with Filter (NPS+f) during its use in a transcarotid stenting procedure. The MICHI NPS+f is an embolic protection device that uses reverse flow to protect the brain during stenting of the Internal Carotid Artery. It is CE marked and is used in routine practice for the purpose of this study.

ELIGIBILITY:
Inclusion and exclusion criteria per CE marked Instructions For Use

Inclusion Criteria:

1. Adequate central venous access
2. Common carotid artery reference diameter of at least 6 mm
3. Carotid bifurcation is a minimum of 5 cm above the clavicle as measured by duplex Doppler ultrasound (DUS) or computerized axial tomography (CT) angiography or magnetic resonance (MR) angiography

Exclusion Criteria:

1. Patients in whom antiplatelet and/or anticoagulation therapy is contraindicated
2. Patients with unresolved bleeding disorders
3. Patients with severe disease of the ipsilateral common carotid artery

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients who are booked for a routine stenting of the Internal Carotid Artery (bifurcation may be involved) using the MICHI(TM) NPS+f System, at vascular surgery departments or interventional radiology departments
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with debris captured in the MICHI(TM) inline filter | During MICHI(TM) NPS+f procedure
  The percentage of patients with any debris captured in the MICHI(TM) inline filter will be calculated

SECONDARY OUTCOMES:
Volume of debris captured in the MICHI(TM) inline filter | During MICHI(TM) NPS+f procedure
  For all patients, where debris is captured in the MICHI(TM) inline filter, the volume of debris will be measured
Histological analysis of debris captured in the MICHI(TM) inline filter | During MICHI(TM) NPS+f procedure
  For all patients, where debris is captured in the MICHI(TM) inline filter, the type of plaque will be determined.

CONTACTS AND LOCATIONS:
Locations (6):
- University Hospital, Ghent, Belgium
- Augusta Krankenhaus, Düsseldorf, Germany
- Spain (4):
  - University Hospital Son Espases, Palma, Mallorca
  - Hospital Vall d'Hebron, Barcelona
  - Hospital Medico Quirurgic, Jaén
  - Complejo Hospitalario de Toledo, Toledo